CLINICAL TRIAL: NCT00522678
Title: A Randomised, Double Blind, Placebo Controlled, Parallel Group, 14 Day Repeat Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled GW685698X Containing Magnesium Stearate in Healthy Subjects
Brief Title: Repeat Dose GW685698X With Magnesium Stearate, Excipient Bridging Study, In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: HZA102928
Record Dates: First submitted 2007-03-07; First posted 2007-08-30 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Healthy Volunteers
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): In Cohort A, subjects will be randomized (3:1) to receive once daily doses of GW685698X 400 microgram (mcg) containing magnesium stearate or placebo via DISKUS, for 14 days.
  Interventions: Drug: GW685698X; Drug: Placebo
- Cohort B (Experimental): In Cohort B, subjects will be randomized (3:1) to receive once daily doses of GW685698X (600 mcg) containing magnesium stearate or placebo via DISKUS, for 14 days.
  Interventions: Drug: GW685698X; Drug: Placebo
- Cohort C (Experimental): InIn Cohort C, subjects will be randomized (3:1) to receive once daily doses of GW685698X (800 mcg) containing magnesium stearate or placebo via DISKUS, for 14 days.
  Interventions: Drug: GW685698X; Drug: Placebo

INTERVENTIONS:
Drug: GW685698X — Subject will receive GW685698X containing magnesium stearate with unit dose strength of 400, 600 and 800 mcg inhaled via DISKUS
Drug: Placebo — Subject will receive Placebo matching GW685698X via DISKUS.

SUMMARY:
GW685698X is a novel glucocorticoid receptor agonist that is being developed as an orally inhaled treatment for asthma. In previous studies inhaled GW685698X was administered as a dry powder containing either lactose alone or lactose and cellobiose octaacetate. However, future dry powder GW685698X formulations will contain lactose and magnesium stearate. This study will be the first administration of this new GW685698X dry powder formulation in man and will provide safety and tolerability data to support the further development of this formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers,
* Aged 18-65
* Male and females (females of non-child bearing potential or who meet the contraception criteria).
* BMI - 19-31 kg/m2

Exclusion Criteria:

* History of breathing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-02-15 (Actual); Primary Completion 2007-04-25 (Actual); Study Completion 2007-04-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Vital signs: systolic and diastolic blood pressure (BP), heart rate (HR) 12-lead ECG including QT, QTc, PR and QRS intervals PEFR Laboratory safety tests (clinical chemistry, haematology, urinalysis) Adverse events | Up to Day 16

SECONDARY OUTCOMES:
Plasma concentrations and pharmacokinetic parameters (AUC, Cmax, t1/2, tmax) for GW685698X on Day 1 and Day 14. Weighted mean serum cortisol, (0-24 h) on Day 14. | Weighted mean serum cortisol, (0-24 h) on Day 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Results for study HZA102928 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/HZA102928?search=study&search_terms=HZA102928#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: HZA102928 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HZA102928 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HZA102928 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HZA102928 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HZA102928 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HZA102928 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HZA102928 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register